CLINICAL TRIAL: NCT03690089
Title: Low-dose Atropine Eye Drops to Reduce Progression of Myopia in Children: a Multi-centre Placebo Controlled Randomised Trial in the United Kingdom
Brief Title: Low-dose Atropine Eye Drops to Reduce Progression of Myopia in Children in the United Kingdom
Acronym: CHAMP-UK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17097AB-AS; 2017-004108-23 (EudraCT Number)
Record Dates: First submitted 2018-08-20; First posted 2018-10-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-masked, placebo-controlled superiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Atropine 0.01%) (Experimental): The intervention group will receive 0.01% atropine sulfate eye drops, administered once daily for two years.
  Interventions: Drug: Atropine Sulfate
- Placebo Group (Placebo Comparator): The control group will receive placebo eye drops, administered once daily for two years.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atropine Sulfate — Atropine sulfate 0.01% eye drops which consist of 10mls of a clear colourless solution of atropine sulfate 0.01% w/v and benzalkonium chloride 0.01% w/v in sterile water.
  Arms: Intervention Group (Atropine 0.01%)
Other: Placebo — Placebo eye drops which consist of 10mls of a clear colourless solution of benzalkonium chloride 0.01% w/v in sterile water.
  Arms: Placebo Group

SUMMARY:
Short-sightedness, also called myopia, makes objects in the distance, such as the television, look blurred. This is caused by the eye growing too long, something that usually happens while children are also getting taller. People with myopia can see better with glasses or contact lenses, but this doesn't stop their eyes continuing to become more short-sighted. The CHAMP UK study is investigating a type of eye drop called atropine that might help to stop myopia getting worse as children get older.

DETAILED DESCRIPTION:
The study hypothesis is that low dose atropine eye drops will reduce the progression of short-sightedness in children compared with placebo eye drops. This is a randomised controlled trial which will be conducted across four Clinical Research Facilities associated with higher education institutions in the UK. It is a double masked trial, that is, neither the participant or the research team will know what treatment the participants are receiving. 289 children aged 6-12 years with short-sightedness will be recruited to the trial. They will be randomly chosen to receive either atropine eye drops or placebo eye drops on a 2:1 basis. Therefore, 193 participants will receive atropine eye drops, 96 participants will receive placebo eye drops.

Potential participants will be referred either by their high street optician or their parents will refer them directly. The study will be advertised on local radio. Potential participants will be invited to attend a baseline screening visit. Written informed consent and written informed assent will be obtained from the parent and child prior to undertaking any assessments. Potential participants will undergo a number of assessments similar to what is conducted by the high street optician or eye clinic to determine if they are eligible to participate. These include: assessment of near and distance vision, reading speed and different measurements of the eye using instruments. An eye drop will be put into each eye for some of these assessments. These drops cause a short-term increase in pupil size, which may last for 12-24 hours, and make close up vision (through their glasses) blurry for up to four hours, and may make them more sensitive to bright light. Participants will also be asked about their quality of life and their daily activities such as screen time, playing outside and reading.

Participants will be instructed in the use of the eye drops. They will put one drop in each eye daily for 24 months. The atropine eye drops contain 0.01% atropine sulphate. Placebo eye drops have been chosen as the comparator group as there is no alternative treatment for this condition. Participants will be given a six month supply of eye drops at each visit (except the last visit at 24 months). This will include seven bottles as each bottle can only be used for 28 days after opening.

Participants will have a further four visits to the research facility for the assessments to be repeated. This will be every six months, therefore five visits in total (baseline, 6 months, 12 months, 18 months and 24 months). It is anticipated that each visit will last approximately 1-2 hours. Children will be offered the opportunity to rest between assessments. At these follow up visits, in addition to the assessments, they will be asked about their tolerability of the eye drops. Also, five years after randomisation, the investigators will post a questionnaire to participants and ask details of any possible complications and adverse events. The investigators will also request information from their optometrist regarding their eye health, distance vision and refractive error data.

The primary outcome is the change in the severity of short-sightedness after 24 months. This will be measured using a machine called an autorefractor.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-12 years (at the time of consenting)
2. Myopia of -0.5D or greater (spherical equivalent refractive error) in both eyes
3. Best-corrected distance visual acuity (BCDVA) 0.20 logMAR or better in both eyes

Exclusion Criteria:

1. Children with other ocular morbidities
2. Myopia of -10D or greater in either eye
3. Astigmatism of 2D or higher in either eye
4. Amblyopia
5. Significant health problems that can compromise the ability to attend research visits or complete the trial
6. Other factors that may compromise the ability to attend the research appointments
7. Parents or children with poor understanding of the English language
8. Children enrolled in other interventional trials
9. Allergy or hypersensitivity to atropine or excipients

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 289 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Spherical equivalent refractive error (i.e. myopia severity) | Baseline - 24-months
  Spherical equivalent refractive error (i.e., myopia severity) of both eyes measured by autorefractor under cycloplegia (adjusted for baseline).

SECONDARY OUTCOMES:
Central axial length | Baseline - 24-months
  Measured using a laser biometer at central fixation conditions.
Best corrected distance visual acuity (BCdVA) (uniocular and binocular) | Baseline - 24-months
  Assessed using the logMAR ETDRS chart. This is a standard letter chart used in research to ensure accuracy and validity of the acuity measurements and has been shown to be repeatable in children.
Near visual acuity (uniocular and binocular) | Baseline - 24-months
  Tested using near logMAR ETDRS at 40 cm.
Reading speed | Baseline - 24-months
  Measured with the Wilkins Rate of Reading test.
Pupil diameter | Baseline - 24-months
  Measured using an autorefractor.
Accommodation | Baseline - 24-months
  Measured prior to the instillation of cycloplegia using the autorefractor. The measures will be taken monocularly in each eye and binocularly (minimum 3 measurements per condition). The accommodation response (accommodation lag) will be determined by calculating the difference between the Accommodation Response (AR = near MSE (autorefractor)) and the Accommodation Stimulus.
Spectacle correction | Baseline - 24-months
  Current spectacle prescription.
Eye drop tolerability | Baseline - 24-months
  Assessed using a 4-point scale to quantify, from the point of view of the participant, (1) local irritation/stinging associated with eye drop instillation; (2) photophobia; and (3) difficulties reading and writing.
Adverse event rates and allergic reactions rates | Baseline - 24-months
  All AEs will be assessed for seriousness, causality, severity and if the adverse event is related to the study drug, for expectedness.
Quality of Life: measured using the EQ-5D-Y | Baseline - 24-months
  The EQ-5D-Y evaluates five dimensions of a child's health (mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy) using three levels (no problems, some problems and a lot of problems). Each response results in a one-digit number, which can be tallied up for the five dimensions. Participants will then indicate their overall health on a visual analogue scale from 0 (worst health you can imagine) to 100 (best health you can imagine).

OTHER OUTCOMES:
Peripheral axial length | Baseline - 24-months
  Measured using a laser biometer at peripheral fixation conditions
Peripheral retinal defocus | Baseline - 24-months
  Measured with the autorefractor at central and peripheral fixation conditions.
Anterior chamber depth | Baseline - 24-months
  Measured with a laser biometer.
Iris colour | Baseline - 24-months
  Measured using a visual grading scale of dark brown, light brown, blue, green, grey.
Height in cms | Baseline - 24-months
  To provide information about the links between the child's development and eye growth and potentially information about lifestyle.
Weight in kgs | Baseline - 24-months
  To provide information about the links between the child's development and eye growth and potentially information about lifestyle.
Hours of outdoor activity | Baseline - 24-months
  Measured using an activities questionnaire.
Ciliary body biometry | Baseline - 24-months
  Measured using anterior-segment OCT (AS-OCT). This will enable changes in lens position and ciliary muscle changes resulting from atropine use to be compared with normal myopic growthChorio-retinal thickness: measured using spectral domain OCT (SR-OCT). This will enable differences in choroidal thickness resulting from atropine use to be compared with normal myopic growth.

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Azuara-Blanco, PhD FRCOphth, Principal Investigator — Queen's University, Belfast
Locations (4):
- United Kingdom (4):
  - Northern Ireland Clinical Research, Belfast
  - Aston University Eye Clinic, Birmingham
  - Anglia Ruskin University Eye Clinic, Cambridge
  - Centre for Living (Glasgow Caledonian University), Glasgow

REFERENCES:
- [Derived] Azuara-Blanco A, Logan N, Strang N, Saunders K, Allen PM, Weir R, Doherty P, Adams C, Gardner E, Hogg R, McFarland M, Preston J, Verghis R, Loughman JJ, Flitcroft I, Mackey DA, Lee SS, Hammond C, Congdon N, Clarke M. Low-dose (0.01%) atropine eye-drops to reduce progression of myopia in children: a multicentre placebo-controlled randomised trial in the UK (CHAMP-UK)-study protocol. Br J Ophthalmol. 2020 Jul;104(7):950-955. doi: 10.1136/bjophthalmol-2019-314819. Epub 2019 Oct 25. PMID 31653669